CLINICAL TRIAL: NCT01237301
Title: Comparison of Clinical Decisions and Outcomes Employing a Treat to Target Design for Subjects With Type 2 Diabetes Randomized to Either SMBG or CGM
Brief Title: Comparing Self Monitored Blood Glucose (SMBG) to Continuous Glucose Monitoring (CGM) in Type 2 Diabetes
Acronym: REACT3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Roche Diagnostics GmbH (Industry); International Diabetes Center at Park Nicollet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04034-10-C
Record Dates: First submitted 2010-11-02; First posted 2010-11-09 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2013-11

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CGM Group (Experimental): Wear an unblinded CGM for 16 weeks. Subjects continued previously started medication regiments for their diabetes. Subjects in this arm were randomized to use real time continuous glucose monitoring (rt CGM).
  Interventions: Device: CGM Group
- SMBG Group (Active Comparator): Use SMBG 4 to 7 times a day for 16 weeks. Subjects continued previously started medication regiments for their diabetes. Subjects in this arm were randomized to use structured self monitoring blood glucose (stSMBG) and periodic, blinded continuous glucose monitoring (CGM).
  Interventions: Device: SMBG Group

INTERVENTIONS:
Device: CGM Group — Using CGM unblinded for 16 weeks versus fingersticks 4 to 7 times a day to evaluate which is more beneficial in type 2 diabetes.
  Other Names: DexCom SevenPlus CGM; AccuChek Aviva blood glucose meter
  Arms: CGM Group
Device: SMBG Group — Fingersticks 4 to 7 times a day to evaluate which is more beneficial in type 2 diabetes. Used CGM blinded once every four weeks.
  Other Names: AccuChek Aviva blood glucose meter; DexCom SevenPlus CGM
  Arms: SMBG Group

SUMMARY:
The purpose of this study is to evaluate the use of SMBG and CGM for clinical decisions related to the management of type 2 diabetes. The secondary objective is to determine the benefit of using CGM for clinical diabetes management decision-making.

DETAILED DESCRIPTION:
This study involves the use of the following 2 glucose monitoring methods to measure your blood sugar (glucose) levels and help manage type 2 diabetes:

1. Self Monitoring Blood Glucose (SMBG): blood glucose is measured 4-7 times each day using finger sticks and an blood glucose meter.
2. Continuous Glucose Monitoring (CGM): blood glucose is measured continuously via the CGM device. This device has been approved for use by the U.S. Food and Drug Administration (FDA).

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 and ≤75 years of age (Upper range to assure dexterity for use of CGM)
* Clinical diagnosis of type 2 diabetes
* HbA1c ≥7.0%
* Diabetes can be treated with any of the following therapies within one month prior to study enrollment: (1) medical nutrition therapy alone or with metformin; (2) sulfonylurea with or without metformin; (3) dipeptidyl peptidase 4 (DPP-4) inhibitor or Glucagon-like peptide-1 (GLP-1) agonist with or without metformin; or insulin with or without metformin.

Exclusion Criteria:

* Treated with Thiazolidinediones (TZD)
* Administered prednisone or cortisone medications in the previous 30 days
* Currently pregnant or planning pregnancy during the study period
* Presence of any severe medical or psychological condition or chronic conditions/infections that in the opinion of the Investigator would compromise the subject's safety or successful participation in the study
* HbA1c <7.0%
* Unable to follow the study protocol
* Unable to speak, read and write in English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2010-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard M. Bergenstal, MD, Principal Investigator — International Diabetes Center at Park Nicollet
Locations (1):
- International Diabetes Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Mazze RS, Strock E, Wesley D, Borgman S, Morgan B, Bergenstal R, Cuddihy R. Characterizing glucose exposure for individuals with normal glucose tolerance using continuous glucose monitoring and ambulatory glucose profile analysis. Diabetes Technol Ther. 2008 Jun;10(3):149-59. doi: 10.1089/dia.2007.0293. PMID 18473688

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period October 29, 2010 through November 25, 2011. Study Location: Clinic
Groups:
- CGM Group: Wear an unblinded CGM for 16 weeks.
  Continuous Glucose Monitoring (CGM) : Using CGM unblinded for 16 weeks versus fingersticks 4 to 7 times a day to evaluate which is more beneficial in type 2 diabetes.
- SMBG Group: Use SMBG 4 to 7 times a day for 16 weeks.
  Continuous Glucose Monitoring (CGM) : Using CGM unblinded for 16 weeks versus fingersticks 4 to 7 times a day to evaluate which is more beneficial in type 2 diabetes.
Period: Overall Study
Arm/Group | CGM Group | SMBG Group
Started | 65 | 59
Completed | 60 | 55
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CGM Group | SMBG Group | Total
Number analyzed (Participants) | 65 | 59 | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 47 | 93
  >=65 years | 19 | 12 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (8.9) | 58.8 (10) | 59 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 32 | 61
  Male | 36 | 27 | 63
Region of Enrollment [Number; unit: participants]
  United States | 65 | 59 | 124

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Hemoglobin A1c
Time Frame: 2 week baseline to 16 week final
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | CGM Group | SMBG Group
Number analyzed (Participants) | 65 | 59
percentage of HbA1c | -1.12 (1.07) | -0.82 (0.91)

2. Secondary Outcome: Glucose Exposure (Area Under the Diurnal Median Curve)
Description: The secondary objective is to determine the incremental benefit of CGM for clinical decision-making by using (area under the diurnal median curve). Data was collected to create the curve at every hour of modal day. Example: hours 1-24 of each day. Modal day reflects 14 days worth of CGM data aggregated into a single 24 hour day graph.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Arm/Group | CGM Group | SMBG Group
Number analyzed (Participants) | 59 | 55
mcg*hr/mL | -615.98 (924.04) | -522.88 (951.43)

3. Secondary Outcome: Percent of Time in Hypoglycemia Range
Description: The secondary objective is to determine the incremental benefit of CGM for clinical decision-making using percent time in hypoglycemia range (< 50 mg/dL). Numerator: amount of time with a value of 49 mg/dL or less. Denominator: total amount of time of CGM measurement.
  CGM used for this study produced measurements once every 15 minutes or 360 times per day.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: % of time in hypoglycemia
Arm/Group | CGM Group | SMBG Group
Number analyzed (Participants) | 59 | 55
% of time in hypoglycemia | -0.42 (1.88) | 0.14 (1.22)

4. Secondary Outcome: Change From Baseline in CGM Glucose Variability
Description: Glucose Variability - Interquartile Range used to determine incremental benefit of CGM for clinical decision making. IQR results reflect the change delta from baseline to 16 weeks. IQR is calculated for each subject at each visit. The change in IQR was calculated as final IQR minus baseline IQR. This measure represents an average of the individual subjects IQR delta (baseline to 16 weeks/final).
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CGM Group | SMBG Group
Number analyzed (Participants) | 59 | 55
mg/dL | -8.36 (15.95) | -5.91 (16.73)

ADVERSE EVENTS:
Time Frame: During the period of the 16 week study.
Description: Review every four weeks of SMBG or CGM data as well as patient reported events at each study visit.
Arm/Group | CGM Group | SMBG Group
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/59
Other Adverse Events (participants affected / at risk) | 1/65 | 1/59
OTHER ADVERSE EVENTS (reported when occurring in more than 0.02% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CGM Group (N=65) | SMBG Group (N=59)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes